CLINICAL TRIAL: NCT07166367
Title: A Phase II Single Arm Trial to Assess the Efficacy of ASLAN001 Plus Capecitabine in Previously Irradiated, Progressing Central Nervous System (CNS) Metastases for HER2 Positive Breast Cancer Patients
Brief Title: Phase II Study to Assess the Efficacy of ASLAN001 Plus Capecitabine in CNS Metastases for HER2+ Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficulty in enrolling patients with the illness under study.
Sponsor: National Cancer Centre, Singapore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ASLAN001-006
Record Dates: First submitted 2025-09-03; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: HER2-positive Breast Cancer
MeSH Terms: interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ASLAN001 and Capecitabine (Experimental)
  Interventions: Drug: ASLAN001; Drug: Capecitabine

INTERVENTIONS:
Drug: ASLAN001 — 400mg of Oral ASLAN001 is administered twice daily, every day of each 21-day cycle
  Other Names: Varlitinib; ARRY-543
Drug: Capecitabine — 1000mg/m^2 of Oral Capecitabine is administered twice daily, on Days 1-14 of a 21-day cycle
  Other Names: Xeloda

SUMMARY:
This study is designed to study the efficacy of ASLAN 001 plus capecitabine for previously irradiated, progressing CNS metastases for HER2+ breast cancer patients.

DETAILED DESCRIPTION:
Brain metastasis in breast cancer (BMBC) has very poor prognosis. The focus for this group of patients is on palliation as well as therapeutics that offer meaningful clinical benefits. Treatment options generally involve local control using either whole brain radiotherapy (WBRT) or neurosurgery/radiosurgery or combination of both. Subsequent to local treatment, systemic control can be re-initiated via systemic chemotherapy/targeted therapies or trial participation.

This is a single arm, single center, phase 2 study. A total of 29 eligible HER2 positive breast cancer patients with irradiated, progressing brain metastasis will be enrolled to receive ASLAN001 400 mg orally BID with capecitabine 1000 mg/m2 orally BID for days 1-14 of a 21-day cycle. Treatment will continue until disease progression or unacceptable toxicity.

Baseline brain imaging using either magnetic resonance imaging (MRI) or computed tomography (CT) scans will be performed; non-brain imaging will also be performed in the same settings. Radiological imaging to assess disease status will be performed at baseline and every 2 cycles until disease progression.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with documented histological confirmation of breast cancer with HER-2 overexpression or gene amplification (immunohistochemistry 3+ or immunohistochemistry 2+ with fluorescent / chromogenic / silver in situ hybridization +) prior to study entry.
2. Patients with HER-2-positive breast cancer with brain metastasis (BMBC) who received either radiosurgery and/or WBRT and progressing in CNS.
3. Presence of more than one radiographically measurable brain metastasis.
4. Patients must complete radiation treatment with either whole brain radiotherapy (WBRT) and/or radiosurgery at least 30 days 30 days prior to study entry. (No washout period for other antineoplastic treatment)
5. Patients must be of legal age of more than 21 years old at the time of written informed consent.
6. Patients of childbearing potential to use adequate contraception prior to, during the study, and 12 weeks after the last dose of therapy.
7. Patients able to understand and willing to sign the informed consent form.
8. Patients with Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
9. Patients with acceptable organ and hematological function:

   1. Hematological function:

      * Absolute neutrophil count ≥1.5 × 10**9/L.
      * Platelet count ≥100 × 10**9/L.
      * Hemoglobin ≥9 g/L.
   2. Renal functions:

      - Serum creatinine ≤1.5 × upper limit of normal (ULN).
   3. Hepatic function:

      * Total bilirubin ≤1.5 × ULN.
      * AST and ALT ≤2.5 × ULN (≤5 × ULN if liver metastases are present).

Exclusion Criteria:

1. Patients with malabsorption syndrome, diseases significantly affecting gastrointestinal function, resection of the stomach or small bowel, or difficulty in swallowing and retaining oral medications.
2. Patients with an uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, unstable angina pectoris, cardiac arrhythmia, diabetes, hypertension, or psychiatric illness/social situations that would limit compliance with study requirements.
3. Patients with any history of other malignancy unless in remission for more than 1 year. (Nonmelanoma skin carcinoma and carcinoma-in-situ of uterine cervix treated with curative intent is not exclusionary).
4. Patients who are pregnant or breast-feeding.
5. Patients who were previously treated with ASLAN001 and/or with lapatinib and/or with capecitabine.
6. Patient with known active infection on hepatitis B and hepatitis C and dihydropyrimidine dehydrogenase (DPD) deficiency. (Screening tests not required.)
7. Patients with non-measurable disease alone (i.e. leptomeningeal disease)
8. Patients who need continuous treatment with proton pump inhibitors during the study period.

Ages: 21 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Females with breast cancer
Enrollment: 3 (Actual)
Dates: Start 2016-08-11 (Actual); Primary Completion 2020-01-14 (Actual); Study Completion 2020-01-14 (Actual)

PRIMARY OUTCOMES:
CNS objective response rate (ORR) based on RANO-BM criteria | From start of treatment to date of best response of Complete Response (CR), Partial Response (PR), or Stable Disease (SD), up to 2 years

SECONDARY OUTCOMES:
Safety/toxicity | The time interval between treatment initiation and progression of disease or death from any cause, up to 2 years
  Events with CTCAE grades of 1 and above.
Clinical benefit rate | 12 weeks from the start of treatment
  The sum of complete response (CR) + partial response (PR) + stable disease (SD) at 12 weeks
Progression free survival | The time interval between treatment initiation and progression of disease or death from any cause, up to 2 years
Overall survival | The time interval between treatment initiation and death from any cause, up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Yoon Sim Yap, Principal Investigator — National Cancer Centre, Singapore
Locations (1):
- National Cancer Centre Singapore, Singapore, Singapore